CLINICAL TRIAL: NCT07323732
Title: A Phase II Study of BIO 300 to Reduce the Toxicity of Thoracic Radiotherapy for Patients With Early-Stage Non-Small Cell Lung Cancer and Interstitial Lung Disease (BREATHE)
Brief Title: A Study of BIO 300 and Thoracic Radiation Therapy in People With Non-Small Cell Lung Cancer and Interstitial Lung Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-310
Record Dates: First submitted 2026-01-06; First posted 2026-01-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: NSCLC; NSCLC, Stage I; NSCLC Stage II; Non Small Cell Lung Cancer; Non-small Cell Lung Cancer Stage I; Non-small Cell Lung Cancer Stage II; Interstitial Lung Disease; Interstitial Lung Disease Due to Connective Tissue Disease (Disorder)
Keywords: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Stage I; Non Small Cell Lung Cancer Stage II; NSCLC; NSCLC Stage I; NSCLC Stage II; Interstitial Lung Disease; Interstitial Lung Disease Due to Connective Tissue Disease (Disorder); Memorial Sloan Kettering Cancer Center; 25-310
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Non-Small Cell Lung Cancer and Interstitial Lung Disease (Experimental): Participants with Non-Small Cell Lung Cancer/NCSLC and Interstitial Lung Disease/ILD
  Interventions: Drug: BIO 300

INTERVENTIONS:
Drug: BIO 300 — The drug product, BIO 300 consists of synthetic genistein

SUMMARY:
The purpose of this study to find out whether giving BIO 300 in combination with thoracic radiation therapy is effective in preventing pneumonitis in people with non-small cell lung cancer (NSCLC) and interstitial lung disease (ILD).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. - Patient age ≥ 18 at time of consent
* Stage I - II NSCLC (as per the American Joint Commission on Cancer (AJCC) 8th edition)

  ° Pathologically proven diagnosis of cancer is strongly recommended but is not required if the risk of biopsy is unacceptable. If pathological evidence is not available, there must be clinical evidence for NSCLC and multidisciplinary consensus for treatment.
* Interstitial Lung Disease diagnosis (one of the below)

  * ILD as diagnosed and managed by a pulmonologist
  * ILD based on diagnostic imaging criteria and abnormal DLCO
  * ILD as a result of connective tissue diseases (e.g., polymyositis/dermatomyositis, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, mixed connective tissue disease)
* ECOG performance status of 0 - 3
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Life expectancy of at least 6 months

Exclusion Criteria:

* Previous thoracic radiation
* History of pneumonectomy
* Major surgical procedure (e.g. intra-cranial, intra-thoracic, intra-abdominal, or intra-pelvic) within 28 days prior to enrollment.
* Severe concurrent illness that may preclude timely completion of thoracic radiation or study procedures
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* ILD exacerbation requiring hospitalization in the last 30 days
* Poorly controlled cardiac arrhythmias not responding to medical therapy or a pacemaker
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential unless they are willing to employ a highly effective non-estrogen based contraception from screening to 30 days after the last dose of BIO 300 or to abstain from sexual intercourse during these time periods.

  1. Effective method of non-estrogen-based contraception: condom and a diaphragm, condom and intrauterine device, condom and Depo-Provera, condom and Nexplanon, or condom and progesterone mini-pill
  2. Women who have been off estrogen contraceptives for a minimum 5 days prior to the first scheduled day of study intervention dosing are eligible.
* Concomitant medications:

  1. Any investigational anticancer therapy.
  2. Planned concurrent chemotherapy or immunotherapy
  3. Biologic drugs targeting the immune system (e.g. TNFα blockers, anakinra, rituximab, abatacept, tocilizumab) planned to be use concurrently with BIO 300

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-01-06 (Estimated); Study Completion 2029-01-06 (Estimated)

PRIMARY OUTCOMES:
Pneumonitis free survival | Up to 36 months
  The primary objective of this study is to assess the improvement in the Grade ≥ 3 pneumonitis free survival in participants with Interstitial Lung Disease/ILD treated with BIO 300 in combination with thoracic radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Narek Shaverdian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org